CLINICAL TRIAL: NCT03158701
Title: Prevelance of Fragmented QRS Complex and Prolonged QT Interval in Cirrhotic Patients and Its Correlation With the Severity of the Disease
Brief Title: Prevelance of Fragmented QRS Complex and Prolonged QT Interval in Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Refaat Edwar Nasrallah, internal medicine resident,Assiut University hospital, Assiut University
Other Study IDs: assiut university 7000
Record Dates: First submitted 2017-05-14; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Liver Cirrhosis
Keywords: evaluation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
.Cardiac affection in liver cirrhosis is a clinical condition characterized by impaired diastolic relaxation and contractility with electrophysiological abnormalities.

.Cirrhotic patients with cardiac abnormality have higher mortality rates compared to patients without cardiac affection.

The suggested pathophysiologic mechanisms of cardiac affection in cirrhotic patients are; alterations in the beta-adrenergic signaling pathway and, myocardial fibrosis formation, sympathetic nervous system activation and changes in ion channels.

.As a component of cardiac involvement in cirrhotic patients fragmented QRS complex and prolongation of the corrected QT interval has been documented in most of the cases with liver cirrhosis (LC) and its prevalence increases with the severity of the disease

DETAILED DESCRIPTION:
.Cardiac affection in liver cirrhosis is a clinical condition characterized by impaired diastolic relaxation and contractility with electrophysiological abnormalities.

.Cirrhotic patients with cardiac abnormality have higher mortality rates compared to patients without cardiac affection.

The suggested pathophysiologic mechanisms of cardiac affection in cirrhotic patients are; alterations in the beta-adrenergic signaling pathway and, myocardial fibrosis formation, sympathetic nervous system activation and changes in ion channels.

.As a component of cardiac involvement in cirrhotic patients fragmented QRS complex and prolongation of the corrected QT interval has been documented in most of the cases with liver cirrhosis (LC) and its prevalence increases with the severity of the disease.

.Fragmented QRS (fQRS) is a convenient marker of myocardial scar evaluated by 12-lead electrocardiogram (ECG) recording. fQRS is defined as additional spikes within the QRS complex. In patients with CAD, fQRS was associated with myocardial scar detected by single photon emission tomography and was a predictor of cardiac events. fQRS was also a predictor of mortality and arrhythmic events in patients with reduced left ventricular function. The usefulness of fQRS for detecting myocardial scar and for identifying high-risk patients has been expanded to various cardiac diseases, such as cardiac cirrhosis, arrhythmogenic right ventricular cardiomyopathy, acute coronary syndrome. fQRS can be caused by zigzag conduction around the scarred myocardium, resulting in multiple spikes within the QRS complex .

ELIGIBILITY:
Inclusion Criteria:

* All cirrhotic patients based on history and clinical diagnosis

Exclusion Criteria:

1. Patients known to be rheumatic heart disease
2. Patients known to be hypertensive
3. patients with documented significant coronary artery disease
4. patients taking drugs that affect QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To evaluate the relationship between the presence of FQRS complex and prolonged QT interval in ECG in cirrhotic patients and its correlation with the severity of the disease according to the pugh-child score.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
the measurement that will be used is the presence of fragmented QRS complex and prolonged QT interval in Electrocardiography in patients with liver cirrhosis | one year
  Primary (main) out come:
  To evaluate the relationship between the presence of FQRS complex and prolonged QT interval in ECG in cirrhotic patients and its correlation with the severity of the disease according to the pugh-child score.

IPD SHARING:
Plan to Share IPD: No